CLINICAL TRIAL: NCT06216496
Title: Evaluation of Amino Acid Metabolism Changes in Participants With Ovarian Cancer by Dynamic Test
Brief Title: Evaluation of Amino Acid Metabolism Changes in Ovarian Cancer
Acronym: AMINOCANCER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC20.038; 2022-A01369-34 (Other: ID/RCB)
Record Dates: First submitted 2023-12-26; First posted 2024-01-22 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2023-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic test (Experimental)
  Interventions: Other: dynamic test for amino acid metabolism

INTERVENTIONS:
Other: dynamic test for amino acid metabolism — Subjects are fasting, and the dynamic test is performed as follows:
  Placement of 1 peripheral venous line (for infusions).
  * H0-H1.5: infusion of a 10% glucose solution at increasing flow rate (3 steps of 30 min each: 0.06g/kg/h then 0.12g/kg/h then 0.25g/kg/h of glucose)
  * H1,5: initial blood sampling (amino acid assay)
  * H1.5-H4.5: infusion of amino acid solution (Aminoven 5%, Fresenius Kabi, Sèvres, France) at constant speed (flow rate 10.5 mg/kg/h of nitrogen or 1.30 ml/kg/H) in Y with glucose infusion (0.25g/kg/h of glucose)
  * H4.5: Final blood sampling (amino acid assay) Each amino acid is plotted as a function of its perfusion rate on the abscissa and its variation in plasma concentration on the ordinate.

SUMMARY:
Ovarian cancer is associated with undernutrition in more than half of all cases. The current management of undernutrition-cachexia in cancer is not specific. It is well recognized that the nutritional support currently offered to cancer patients is not effective in combating cachexia, which progresses inexorably, leading to the patient's death. It is therefore necessary to offer specific and adapted care, in particular by optimizing the quality of nitrogen intake. To achieve this, the investigators first need to define the specific amino acid requirements of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of high-grade serous ovarian cancer not immediately resectable (stage III or IVa) managed at Grenoble Alpes University Hospital.
* Affiliation to the French social security system.
* Able to understand and follow the instructions necessary for the conduct of the trial, and having given written consent for the study.

Exclusion Criteria:

* Significant active comorbidity requiring long-term drug treatment (e.g. organ failure, diabetes) or history of pathology likely to impact amino acid metabolism (e.g. urea or homocysteine cycle abnormalities, tyrosinemia, alkaptonuria, hyperprolinemia, organic aciduria).
* vegetarian or vegan diet
* difficult venous access
* Persons covered by articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons: pregnant women, parturients, nursing mothers, persons deprived of their liberty by judicial or administrative decision, persons subject to a legal protection measure).
* Subject receiving more than 4,500 euros in compensation for participation in other research involving the human body in the 12 months preceding this study.
* Significant biological abnormalities (not explained by the underlying pathology for women with ovarian cancer)
* Liver metastases

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
metabolism of each amino acid, in women with non-immediately resectable ovarian cancer (with or without peritoneal metastases) of high-grade serous type. | 270 minutes
  degree of consumption of each amino acid estimated by the difference in plasma concentration in µmol/L measured after 90 minutes (H 1.5) and 270 minutes (H 4.5) of perfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: Undecided